CLINICAL TRIAL: NCT02387827
Title: Comparing of Long Bout and Short Bouts of Similar Volume of Walking in Obese on Weight Loss During a Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-104
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Overweight
Keywords: long bout physical activity; short bout physical activity; Caloric Restriction
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet+ short -term physical activity (DST) (Experimental)
  Interventions: Behavioral: Diet+ short term versus long -term physical activity
- Diet+ long -term physical activity (DLT) (Experimental)
  Interventions: Behavioral: Diet+ short term versus long -term physical activity

INTERVENTIONS:
Behavioral: Diet+ short term versus long -term physical activity

SUMMARY:
The purpose of this present study is to determine if a daily walking program of 50 continuous minutes (long bout) or two 25-minute bouts (short bouts) in similar volume on body weight, abdominal fat mass deposition and cardiometabolic measures in overweight and obese women receiving a low calorie diet for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) between 27-35 kg/ m².
* were sedentary (reported exercising <20 min/d for the previous 6 month) and healthy
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
weight loss | 24 weeks
Body mass index reduction | 24 weeks

SECONDARY OUTCOMES:
waist circumference | 24 weeks
Fasting plasma glucose level | 24 weeks
lipid profiles | 24 weeks
Insulin resistance (HOMA) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NovinDiet Clinic, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Madjd A, Taylor MA, Delavari A, Malekzadeh R, Macdonald IA, Farshchi HR. Effect of a Long Bout Versus Short Bouts of Walking on Weight Loss During a Weight-Loss Diet: A Randomized Trial. Obesity (Silver Spring). 2019 Apr;27(4):551-558. doi: 10.1002/oby.22416. Epub 2019 Feb 9. PMID 30737894